CLINICAL TRIAL: NCT01389973
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Study Evaluating the Efficacy and Safety of Ustekinumab in Subjects With Primary Biliary Cirrhosis Who Had an Inadequate Response to Ursodeoxycholic Acid (UDCA)
Brief Title: A Study of Efficacy and Safety of Ustekinumab in Patients With Primary Biliary Cirrhosis (PBC) Who Had an Inadequate Response to Ursodeoxycholic Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR018748; CNTO1275PBC2001 (Other: Janssen Research & Development, LLC); 2011-000554-31 (EudraCT Number)
Record Dates: First submitted 2011-07-07; First posted 2011-07-08 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Diseases [C] - Digestive System Diseases [C06]; primary biliary cirrhosis; ursodeoxycholic acid (UDCA); STELARA; ustekinumab
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Open-label: ustekinumab 90 mg (Experimental)
  Interventions: Drug: ustekinumab 90 mg
- Double-blind: ustekinumab 45 mg (Experimental)
  Interventions: Drug: ustekinumab 45 mg
- Double-blind: ustekinumab 90 mg (Experimental)
  Interventions: Drug: ustekinumab 90 mg
- Double-blind: ustekinumb 180 mg (Experimental)
  Interventions: Drug: ustekinumab 180 mg
- Double-blind: placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ustekinumab 90 mg — Subcutaneous injections of ustekinumb 90 mg at Weeks 0 and 4 and every 8 weeks until the dose for the Long-Term Extension has been selected then every 8 weeks through Week 196 with the selected dose.
  Arms: Double-blind: ustekinumab 90 mg; Open-label: ustekinumab 90 mg
Drug: ustekinumab 45 mg — Subcutaneous injections of ustekinumb 45 mg at Weeks 0 and 4 and every 8 weeks until the dose for the Long-Term Extension has been selected then every 8 weeks through Week 196 with the selected dose.
  Arms: Double-blind: ustekinumab 45 mg
Drug: ustekinumab 180 mg — Subcutaneous injections of ustekinumb 180 mg at Weeks 0 and 4 and every 8 weeks until the dose for the Long-Term Extension has been selected then every 8 weeks through Week 196 with the selected dose.
  Arms: Double-blind: ustekinumb 180 mg
Drug: Placebo — Subcutaneous injections of placebo at Weeks 0 and 4 and every 8 weeks until the dose for the Long-Term Extension has been selected then every 8 weeks through Week 196 with the selected dose.
  Arms: Double-blind: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ustekinumab in patients with primary biliary cirrhosis who had an inadequate response to ursodeoxycholic acid.

DETAILED DESCRIPTION:
This is a multi-center, randomized (treatment will be assigned by chance), placebo-controlled (an inactive substance will be compared with the test drug to see whether the drug has a real effect), parallel-group (two or more groups of patients will receive different treatments) study that will consist of two parts. Part 1 will be an open-label (all participants will know the identity of the treatment) proof-of-concept study. Part 2 will be contingent on the results of Part 1 and will be double-blind (investigators and patients will not know what treatment is being given) and will evaluate the efficacy and safety of ustekinumab in patients with primary biliary cirrhosis (PBC) who had an inadequate response to ursodeoxycholic acid. The duration of participation in the study for an individual participant may be up to 216 weeks. Patient safety will be monitored. Part 1: ustekinumab, 90mg subcutaneous (SC) at Weeks 0 and 4 and every 8 weeks through Week 20; Part 2: Depending on Part 1 results, either (ustekinumab 90mg or 45mg or placebo) or (ustekinumab 90mg or 180mg or placebo) SC at Weeks 0 and 4 and every 8 weeks through Week 20; Long-term Extension (including Part 1 and Part 2): beginning at Week 28, every 8 weeks with initially assigned dose until the extension dose has been selected; then every 8 weeks through Week 196 with the selected dose.

ELIGIBILITY:
Inclusion Criteria:

* Have proven or are likely to have Primary Biliary Cirrhosis (PBC)
* Be on a stable dose of ursodeoxycholic acid for at least 6 months prior to Week 0
* Have screening alkaline phosphatase (ALP) level > 1.67 ULN (the upper limit of normal)
* Have screening laboratory test results within protocol-specified limits
* Have no history of latent or active tuberculosis (TB) prior to screening and no signs or symptoms suggestive of active TB upon medical history and/or physical examination.

Exclusion Criteria:

* Has history of gastrointestinal bleeding, secondary to portal hypertension, hepatic encephalopathy, or ascites requiring treatment with diuretics
* Has a screening direct bilirubin > 1.0 mg/dL
* Has a previous liver histology with a diagnosis of steatohepatitis or has a high risk of nonalcoholic steatohepatitis
* Has a previous liver histology with a diagnosis of chronic autoimmune hepatitis or has a high risk of autoimmune hepatitis overlap syndrome
* Testing positive for surface antigen (HBsAg+), regardless of the results of other hepatitis B tests
* Have used colchicine, methotrexate (MTX), azathioprine (AZA), or systemic corticosteroids within 3 months prior to the first administration of study drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- United States (6):
  - Jacksonville, Florida
  - Miami, Florida
  - Naples, Florida
  - Tupelo, Mississippi
  - New York, New York
  - Houston, Texas
- Canada (4):
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Derived] Mousa HS, Lleo A, Invernizzi P, Bowlus CL, Gershwin ME. Advances in pharmacotherapy for primary biliary cirrhosis. Expert Opin Pharmacother. 2015 Apr;16(5):633-43. doi: 10.1517/14656566.2015.998650. Epub 2014 Dec 29. PMID 25543678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study had 2 parts, Part 1 (proof of concept) and Part 2. As per the study design, the study was considered completed after part 1 and part 2 was not initiated. Results shown below are for Part 1 of the study.
Groups:
- Open-label: Ustekinumab 90 mg: In proof of concept phase of Part 1, participants received ustekinumab 90 milligram (mg) subcutaneously at Week 0, 4 and thereafter every 8 weeks through Week 20. Eligible participants entered long-term extension which began at Week 28 and continued through Week 216.
Period: Overall Study
Arm/Group | Open-label: Ustekinumab 90 mg
Started | 20
Completed | 0
Not Completed | 20
Not completed — Lost to Follow-up | 1
Not completed — Trial Stopped by Sponsor | 9
Not completed — Other | 10

BASELINE CHARACTERISTICS:
Population: Efficacy analysis set included all participants who received at least 1 administration of ustekinumab (full or partial).
Arm/Group | Open-label: Ustekinumab 90 mg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Alkaline Phosphatase (ALP) Response at Week 12
Description: The ALP response was defined as a greater than 40 percent (%) decrease from Baseline in ALP concentration at Week 12.
Time Frame: Week 12
Population: Efficacy analysis set included all participants who received at least 1 administration of ustekinumab (full or partial).
Measure: Number; unit: participants
Arm/Group | Open-label: Ustekinumab 90 mg
Number analyzed (Participants) | 20
participants | 0

2. Secondary Outcome: Part 1: Number of Participants With ALP Response at Week 28
Time Frame: Week 28
Population: Efficacy analysis set included all participants who received at least 1 administration of ustekinumab (full or partial).
Measure: Number; unit: participants
Arm/Group | Open-label: Ustekinumab 90 mg
Number analyzed (Participants) | 20
participants | 0

3. Secondary Outcome: Part 1: Number of Participants With ALP Remission at Week 28
Description: ALP remission is defined as either normalization of ALP (for participants with baseline ALP between 1.67*and 2.8* upper limit of normal [ULN] or an ALP less than [˂]1.67*ULN [for participants with baseline ALP greater than {˃} 2.8* ULN]). ALP levels above 1.67* ULN level were associated with an increased rate of disease progression.
Time Frame: Week 28
Population: Efficacy analysis set included all participants who received at least 1 administration of ustekinumab (full or partial).
Measure: Number; unit: participants
Arm/Group | Open-label: Ustekinumab 90 mg
Number analyzed (Participants) | 20
participants | 0

4. Secondary Outcome: Part 1: Percent Change From Baseline in ALP Concentration at Week 28
Time Frame: Baseline and Week 28
Population: Efficacy analysis set included all participants who received at least 1 administration of ustekinumab (full or partial).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Open-label: Ustekinumab 90 mg
Number analyzed (Participants) | 20
percent change | -11.25 (17.462)

5. Secondary Outcome: Part 1: Percent Change From Baseline in Alanine Aminotransferase, Aspartate Aminotransferase, and Bilirubin Concentration at Week 28
Time Frame: Baseline and Week 28
Population: Efficacy analysis set included all participants who received at least 1 administration of ustekinumab (full or partial). "N" (number of participants analyzed) signifies participants who were evalubale for this outcome measure. "n" signifies participants who were evalubale for each specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Open-label: Ustekinumab 90 mg
Number analyzed (Participants) | 18
percent change
  Alanine Aminotransferase (n=18) | -9.21 (32.362)
  Aspartate Aminotransferase (n=18) | -7.22 (27.188)
  Bilirubin (n=3) | -4.61 (14.183)

ADVERSE EVENTS:
Time Frame: Week 0 up to final safety visit in Part 1
Arm/Group | Open-label: Ustekinumab 90 mg
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label: Ustekinumab 90 mg (N=20)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label: Ustekinumab 90 mg (N=20)
Fatigue (General disorders) | 8
Feeling abnormal (General disorders) | 1
Injection site bruising (General disorders) | 1
Injection site erythema (General disorders) | 1
Pyrexia (General disorders) | 1
Urinary tract infection (Infections and infestations) | 4
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Salivary gland enlargement (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 5
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Weight decreased (Investigations) | 1
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Based on the efficacy results of Part 1, Part 2 of the study was not initiated and as per the study design, the study was considered completed after part 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less